CLINICAL TRIAL: NCT05776953
Title: Evaluation of the Effects of Ketorolac 15mg IV Versus 30mg IV on Duration of Analgesia in Patients Who Present to the Emergency Department With Renal Colic
Brief Title: Evaluation of the Effects of Ketorolac Dose on Duration of Analgesia in Emergency Department (ED) Renal Colic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro2022-0546
Record Dates: First submitted 2023-02-27; First posted 2023-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Renal Colic; Flank Pain; Emergencies; Analgesia
MeSH Terms: conditions — Renal Colic; Flank Pain; Emergencies; Agnosia | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient, treating provider, and the investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 15mg IV Ketorolac (Active Comparator): Patients will be randomized to 15mg IV ketorolac
  Interventions: Drug: Ketorolac
- 30mg IV Ketorolac (Active Comparator): Patients will be randomized to 30mg IV ketorolac
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — IV Ketorolac for pain

SUMMARY:
This is a prospective interventional study examining the effect of ketorolac at doses of 15mg versus 30 mg for duration of analgesia in emergency department patients with suspected renal colic.

DETAILED DESCRIPTION:
Pain is a common emergency department complaint. With various types of analgesics available, the optimal drug is one that provides adequate pain management with minimal side effects. The goal is to effectively treat the patient while maintaining adequate flow in the emergency department. In cases of moderate to severe pain in emergency departments, opioids have been the gold standard.1 Opiates, such as morphine, are associated with side effects that can be distressing to the patient, as well as, costly to the department. Prescribing opiates includes a reluctance in administering sufficient opioid dosing due to fear of tolerance and dependency.2

It has been demonstrated in other studies that the standard dosing of ketorolac is higher than needed to achieve analgesia but have failed to show to what duration of time analgesia is maintained between the dosages. The study will compare the analgesic efficacy of two doses of intravenous ketorolac (15mg and 30mg) for acute flank pain in the Emergency Department (ED), such as renal colic, and how efficacious the pain was controlled at 120 minutes or upon discharge. Motov et al evaluated the effectiveness of ketorolac in moderate to severe pain with a primary endpoint of 30 minutes, however the peak onset of ketorolac is 120 to 180 minutes.

Our study may further investigate the ceiling dose of intravenous ketorolac. The primary outcome of both Motov et al and Eidinejad et al was pain reduction 30 minutes after ketorolac administration.3,4 These studies differed in the aspect that Eidinejad et al study examined pain reduction up to 60 minutes, while Motov et al observed up to 120 minutes after administration of ketorolac.3,4 Ketorolac has a peak time of onset at 2 to 4 hours. These studies are not observing ketorolac at its optimal analgesic potency. Therefore, a study is proposed to compare 15 mg vs 30 mg intravenous ketorolac with the primary outcome being pain reduction in renal colic at 120 minutes. Nephrolithiasis and ureterolithiasis are the most common diagnoses in the emergency department for which ketorolac is prescribed.5 This study may further evaluate optimal intravenous ketorolac dosing in pathology it is known to be the most advantageous.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they present to the Emergency Department with (all of the following):

* Adult emergency department patients < 65 years old
* One or more of the following common ED chief complaints associated with the suspected diagnosis of renal colic. These chief complaints include but are not limited to: flank pain, back pain, abdominal pain, left and/or right lower quadrant pain, and/or pelvic pain
* Pain score of 4 or greater on the 0-10 NRS
* Determination of treatment with IV ketorolac

Exclusion Criteria:

Patients will be excluded if any of the following apply:

* Allergy to ketorolac
* Pregnant patients
* Previously received analgesic medications within 4 hours prior to administration of ketorolac in our ED
* Known or stated history of renal insufficiency
* Body weight < 50 kg
* Age greater than 65 years
* Patients that do no read/write Spanish or English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain scale post ketorolac administration | At 120 minutes (+/-10 minutes) from medication administration
  This study may prospectively compare the mean Numerical Rating Scale (NRS) pain score reduction of 15 mg versus 30 mg of intravenous (IV) ketorolac at 120 minutes after administration to treat renal colic in the emergency department. The scale ranges from 0 to 10 with 0 being "no pain" and 10 being "very much pain".

SECONDARY OUTCOMES:
Change in pain scale post ketorolac administration at different time points | At 90 minutes (+/-10 minutes) from medication administration
  This study may also determine the mean NRS pain score reduction at different time points (90 minutes, 150 minutes, and 180 minutes) after IV ketorolac administration. The scale ranges from 0 to 10 with 0 being "no pain" and 10 being "very much pain".
Change in pain scale post ketorolac administration at different time points | At 150 minutes (+/-10 minutes) from medication administration
  This study may also determine the mean NRS pain score reduction at different time points (90 minutes, 150 minutes, and 180 minutes) after IV ketorolac administration. The scale ranges from 0 to 10 with 0 being "no pain" and 10 being "very much pain".
Change in pain scale post ketorolac administration at different time points | At 180 minutes (+/-10 minutes) from medication administration
  This study may also determine the mean NRS pain score reduction at different time points (90 minutes, 150 minutes, and 180 minutes) after IV ketorolac administration. The scale ranges from 0 to 10 with 0 being "no pain" and 10 being "very much pain".
Need for additional rescue analgesia | At 120 minutes from medication administration
  Study may also examine the number of patients requesting rescue analgesia within two hours of ketorolac administration (yes vs. no)
Type of additional rescue analgesia needed | At 120 minutes from medication administration
  For the patients who need additional pain medication, we will collect the type of medication provided.
Dose of additional rescue analgesia needed | At 120 minutes from medication administration
  For the patients who need additional pain medication, we will collect the dose of medication provided.

CONTACTS AND LOCATIONS:
Overall Officials: Biren Bhatt, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univarsity medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelinek GA. Ketorolac versus morphine for severe pain. Ketorolac is more effective, cheaper, and has fewer side effects. BMJ. 2000 Nov 18;321(7271):1236-7. doi: 10.1136/bmj.321.7271.1236. No abstract available. PMID 11082068
- [Background] Catapano MS. The analgesic efficacy of ketorolac for acute pain. J Emerg Med. 1996 Jan-Feb;14(1):67-75. doi: 10.1016/0736-4679(95)02052-7. PMID 8655940
- [Background] Motov S, Yasavolian M, Likourezos A, Pushkar I, Hossain R, Drapkin J, Cohen V, Filk N, Smith A, Huang F, Rockoff B, Homel P, Fromm C. Comparison of Intravenous Ketorolac at Three Single-Dose Regimens for Treating Acute Pain in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2017 Aug;70(2):177-184. doi: 10.1016/j.annemergmed.2016.10.014. Epub 2016 Dec 16. PMID 27993418
- [Background] Eidinejad L, Bahreini M, Ahmadi A, Yazdchi M, Thiruganasambandamoorthy V, Mirfazaelian H. Comparison of intravenous ketorolac at three doses for treating renal colic in the emergency department: A noninferiority randomized controlled trial. Acad Emerg Med. 2021 Jul;28(7):768-775. doi: 10.1111/acem.14202. Epub 2021 Feb 17. PMID 33370510
- [Background] Soleyman-Zomalan E, Motov S, Likourezos A, Cohen V, Pushkar I, Fromm C. Patterns of Ketorolac dosing by emergency physicians. World J Emerg Med. 2017;8(1):43-46. doi: 10.5847/wjem.j.1920-8642.2017.01.008. PMID 28123620